CLINICAL TRIAL: NCT03176251
Title: Gamification of a Virtual-reality Simulation Curriculum in Endoscopy: Impact on Clinical Performance
Brief Title: Applying Gamification to Postgraduate Endoscopic Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Unity Health Toronto (Other)
Responsible Party: Principal Investigator, Samir Grover, Dr. Samir C. Grover, MD, MEd, FRCPC, Unity Health Toronto
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 17-092
Record Dates: First submitted 2017-06-01; First posted 2017-06-05 (Actual); Last update posted 2021-01-14 (Actual); Status verified 2021-01

CONDITIONS: Endoscopy; Gamification; Simulation

STUDY DESIGN:
Intervention Model Description: Randomized, two-arm, single-blinded
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group: Conventional Training Group (Active Comparator): This group will receive 4 hours of didactic and hands-on sessions on colonoscopy theory and non-technical skills. Participants will also watch a video that demonstrates an ideal endoscopic procedure. After each didactic session, a short multiple-choice questionnaire based on the topics covered in that session will be administered. In addition to didactic training, the control group will be given six hours of expert-assisted instruction on low-fidelity (1 hour) and high-fidelity (5 hours) colonoscopy simulators. Six modules of increasing difficulty in colonoscopy will be taught using one-on-one feedback from an expert academic endoscopist. The endoscopy instructor will demonstrate techniques and provide feedback. During training on the high-fidelity simulator, the last two hours will take the form of the integrated scenario, which will feature a standardized patient (SP) and standardized nurse (SN). Feedback will be given after each integrated scenario by the instructor.
  Interventions: Other: Gamified-Integrated Curriculum
- Intervention Group: Gamified-Integrated Curriculum (GIC) (Experimental): The intervention group will receive the same core training as the control group with additional elements of gamification: leaderboards and badges. First, leaderboards will be used to track and rank participants' performances. This will be done through an anonymized ID tag that allows a participant to identify only their position on the leaderboard. This leaderboard will include 4 components: non-technical skills, technical skills, cognitive skills, and overall ranking. Scores will be aggregated only from participants training on the same days. The leaderboard will be displayed on a central laptop and/or TV screen and will be accessible at any time throughout the day. Second, participants in the GIC group will have the opportunity to be rewarded for their performances using achievement badges which are visual cues to the player that he or she has achieved something. Awards will be given to participants at the top of the leaderboard and with the most badges.
  Interventions: Other: Gamified-Integrated Curriculum

INTERVENTIONS:
Other: Gamified-Integrated Curriculum — The experimental group will receive identical training compared to the control group, with the additional incorporation of several elements of gamification, as outlined in the Arm/Group descriptions.

SUMMARY:
Simulation-based training curricula for gastrointestinal endoscopy have been developed and have been shown to be effective. It is possible that these curricula may be further improved. Gamification, the application of game-design principles to non-game contexts, has been shown to improve learning and skill performance in medical education. In gastrointestinal endoscopy, however, no dedicated curricula have been developed using gamification principles. We aim to evaluate the impact of applying gamification to a curriculum using SBT in endoscopy on clinical performance, compared to an identical curriculum without gamification. 36 novice endoscopists from the general surgery and gastroenterology programs at the University of Toronto will be recruited. Participants will be randomized into two groups: the Conventional Training Curriculum (CTC) Group, in which participants will receive 6 hours of training on a simulator augmented with expert feedback and interlaced with 4 hours of didactic training on the theory of colonoscopy; and the Gamified Integrated Curriculum (GIC) Group, in which participants will receive the same curriculum, using the following applications of gamified learning: a leaderboard of participant performances; badges for achievement of training landmarks; and rewards for top performance. Participants will be trained to perform colonoscopies progressively moving from a low to high complexity simulators, starting with the bench-top model (1 hour) and then moving to the EndoVR® virtual reality (VR) gastroenterology simulator (5 hours). Performance will be assessed at three points: prior to training (pre-test), immediately after training (acquisition post-test) and 4-6 weeks after training (retention test). Assessment will take place on the simulator at all three time points and during two live colonoscopies at the retention test. The primary outcome measure will be the difference in clinical colonoscopy performance between the two training groups, as assessed by the Joint Advisory Group for GI Endoscopy Direct Observation of Procedural Skills (JAG/DOPS). We aim to have data collection finished by 2018. Our results have the potential to improve existing curricula for training in colonoscopy. Moreover, the development of a gamified curriculum in procedural skills may have applicability to other specialities, such as general surgery and anesthesiology.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be novice endoscopists enrolled in general surgery, adult gastroenterology and pediatric gastroenterology programs at the University of Toronto

Exclusion Criteria:

* Participants will be excluded if they have performed 25 or more real or simulated endoscopic procedures

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2019-08-30 (Actual); Study Completion 2019-08-30 (Actual)

PRIMARY OUTCOMES:
Performance on a clinical colonoscopy | 4-6 weeks post-intervention
  Difference between the control and intervention groups during two clinical colonoscopies as assessed by two independent, blinded, expert endoscopists using the Joint Advisory Group for GI Endoscopy Direct Observation of Procedural Skills (JAG/DOPS)

SECONDARY OUTCOMES:
Procedural Knowledge | Pre-intervention and immediate post-intervention
  Differences between the two groups with respect to procedural knowledge as assessed by multiple-choice questionnaires
Non-technical performance | 4-6 weeks post-intervention
  Differences between the two groups with respect to non-technical performance during clinical colonoscopies and an integrated scenario format test 4-6 weeks after training, as assessed by the modified objective structured assessment of nontechnical skills (M-OSANTS)
Patient comfort | 4-6 weeks post-intervention
  Differences between the two groups with respect to patient comfort during the clinical colonoscopies, as assessed by the Nurse-Assessed Patient Comfort Score (NAPCOMS)
Participant self-efficacy | Pre-intervention, immediate post-intervention, and 4-6 weeks post-intervention
  Differences between the two groups with respect to participant self-efficacy, as measured by an adapted scale based on the General Self-Efficacy Scale
Cognitive load | Pre-intervention, immediate post-intervention, and 4-6 weeks post-intervention
  Differences between the two groups with respect to cognitive load, as measured by the Cognitive Load Scale for Colonoscopy
Technical performance | Immediate post-intervention and 4-6 weeks post-intervention
  Difference between the two groups with respect to technical performance on a VR simulated colonoscopies as assessed through the JAG/DOPS
Participant competitiveness | Pre-intervention
  Difference between the two groups with respect to competitiveness as measured using the Revised Competitiveness Index

CONTACTS AND LOCATIONS:
Locations (1):
- St. Michael's Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Scaffidi MA, Khan R, Walsh CM, Pearl M, Winger K, Kalaichandran R, Lin P, Grover SC. Protocol for a randomised trial evaluating the effect of applying gamification to simulation-based endoscopy training. BMJ Open. 2019 Feb 24;9(2):e024134. doi: 10.1136/bmjopen-2018-024134. PMID 30804029